CLINICAL TRIAL: NCT03084380
Title: Phase I Trial of Anti-GPC3 Chimeric T Cells for Subjects With GPC3-Positive Advanced Hepatocellular Carcinoma
Brief Title: Anti-GPC3 CAR-T for Treating GPC3-positive Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Secretary of research, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPC3CAR
Record Dates: First submitted 2017-03-05; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-GPC3 CAR-T (Experimental): Transcatheter arterial chemoembolization (TACE) combine with GPC3-CART infusion
  Interventions: Biological: Retroviral vector-transduced autologous T cells to express anti-GPC3 CARs; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Retroviral vector-transduced autologous T cells to express anti-GPC3 CARs — transcatheter arterial chemoembolization + CAR-T infusion
Drug: Fludarabine — Fludarabine will be administered at dose of 25mg/m2/d
Drug: Cyclophosphamide — Cyclophosphamide will be administered at dose of 40mg/kg for 1 day and then fludarabine will be given for the next 5 days and then the T cells will be administered

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of anti-GPC3 scFv-41BB-CD3ζ-tEGFR chimeric antigen receptor (CAR)-modified T (CAR-T) cells in treating patients with GPC3-positive advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Primary Objectives:

1. To evaluate the safety of intravenous administration of the anti-GPC3 CAR-T cells in patients with HCC or lung squamous cell carcinoma
2. To access the safety of anti-GPC3 CAR-T cells in HCC patients through catheter injection

Secondary Objectives:

1. To evaluate the efficacy of anti-GPC3 CAR-T cells in patients with advanced HCC or lung squamous cell carcinoma
2. To monitor the serum cytokine and expression level of tumor markers such as AFP, CEA and GPC3
3. To assess the persistence in peripheral blood and intratumoral infiltration of anti-GPC3 CAR-T cells

ELIGIBILITY:
Inclusion Criteria:

* Expected to survive more than 3 months
* PS 0-2
* Immunohistochemistry was confirmed to be GPC3 positive hepatocellular carcinoma
* Patients with no ability to receive TACE combined with sorafenib
* WBC>3.5×1e+9/L,Hb>90g/L,PLT>75×1e+9/L
* HBV DNA copy number less than 100/ml
* ALT≤5ULN, AST≤5ULN, TB≤1.5ULN, ALB≥35g/L
* Understand this test and have signed informed consent

Exclusion Criteria:

* Hepatic encephalopathy, autoimmune diseases, or any uncontrolled active disease that hinders participation in the trial
* Decompensated liver cirrhosis, liver function Child-pugh C grade
* Portal vein tumor thrombus, arterial portal fistula, hepatic arteriovenous
* Long-term use of immunosuppressive agents after organ transplantation
* Screening indicated that the target cell transfection rate was less than 30%
* Invasive pulmonary embolism, deep venous thrombosis, or other major arterial / venous thromboembolic events occurred 30 days or 30 days prior to randomization
* Subjects had an active or uncontrollable infection requiring systemic therapy 14 days or 14 days prior to randomization
* Pregnant or lactating subjects
* In the opinion of the investigator, the presence of a medical history or a history of mental state may increase the number of subjects associated with the risk factors associated with the study or study drug administration
* Subjects who have signed a written consent or who are in compliance with the study procedure; or who are unwilling or unable to comply with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 4 weeks
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0

SECONDARY OUTCOMES:
Efficacy: Overall complete remission rate defined by the standard response criteria | 8 weeks
  Overall complete remission rate defined by the standard response criteria
Persistence: Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes